CLINICAL TRIAL: NCT01377025
Title: A Randomized Discontinuation, Blinded, Placebo-Controlled Phase II Study of Sorafenib in Patients With Chemonaive Metastatic Uveal Melanoma
Brief Title: A Study of Sorafenib in Patients With Chemonaive Metastatic Uveal Melanoma
Acronym: STREAM
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Prof. Dr. med. Max. E. Scheulen (Other)
Collaborators: ClinAssess GmbH (Industry)
Responsible Party: Sponsor-Investigator, Prof. Dr. med. Max. E. Scheulen, Prof,. Dr. med., University Hospital, Essen
Organization: University Hospital, Essen (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STREAM; 2010-022687-12 (EudraCT Number)
Record Dates: First submitted 2011-06-14; First posted 2011-06-20 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Uveal Melanoma
MeSH Terms: conditions — Uveal Melanoma | interventions — Sorafenib

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Sorafenib blinded Phase (Experimental): 400 mg Sorafenib bid until PD
  Interventions: Drug: Sorafenib
- Placebo blinded Phase (Placebo Comparator): Two tbl. in the morning and two tbl. in teh evening until PD
  Interventions: Drug: Placebo
- Sorafenib Open Phase (Experimental): 400 mg Sorafenib bid until PD
  Interventions: Drug: Sorafenib

INTERVENTIONS:
Drug: Placebo — two tablets in the morning and two in the evening.
  Arms: Placebo blinded Phase
Drug: Sorafenib — 400 mg Sorafenib bid until PD if staging after Run-In was PR or CR
  Arms: Sorafenib Open Phase
Drug: Sorafenib — 400 mg Sorafenib bid until PD if staging after Run-In was SD
  Arms: Sorafenib blinded Phase

SUMMARY:
Uveal melanoma is the most common primary intra-ocular malignancy in adults with an incidence of 0.6 - 0.7 per 100,000 per year.

Prognosis of metastatic uveal melanoma is poor. In retrospective analyses a median survival time after detection of metastases of 5 months (Flaherty et al, 1998) and 7 months (Kath et al, 1993) was reported. For patients receiving no treatment reported median survival was 2.0 months compared with 5.2 months for those receiving treatment for metastases (Gragoudas et al, 1991).

Up to now there is no established treatment of metastatic uveal melanoma. Some therapeutic approaches with locoregional treatment or systemic chemotherapy have been undertaken:

In case of metastatic disease which is confined to the liver in about 85% of patients with uveal melanoma surgical resection led to a median survival of 14 months (Mariani et al, 2009) or 19 months and a 5-year survival rate of 22% in a selected patient population (Adam et al, 2006).

As locoregional treatment option treatment with fotemustine via direct intra-arterial hepatic infusion was investigated and led to a median survival of 15 months (Peters et al, 2006). This was not a randomized trial, but a report on 101 consecutive treated patients. Additional debulking surgery was performed whenever feasible.

A randomized phase III trial comparing intra-arterial hepatic fotemustine administration with intravenous systemic fotemustine and overall survival as primary endpoint is still ongoing (EORTC 18021).

Thus, no systemic chemotherapy is approved for metastatic uveal melanoma. Although no specific genes have been linked to the pathogenesis of uveal melanoma, preclinical studies suggest potential benefit of inhibitors of Bcl-2, ubiquitin-proteasome, histone deactylase, mitogen-activated protein kinase and phosphatidylinositol-3-kinase-AKT pathways, and receptor tyrosine kinases.

Thus, sorafenib as inhibitor of b-Raf and Raf-1 (c-Raf or c-Raf-1), pro-angiogenic vascular endothelial growth factor receptor (VEGFR), and platelet-derived growth factor receptor (PDGFR) may potentially lead to a benefit for patients with metastatic uveal melanoma in terms of disease control and prolongation of survival.

DETAILED DESCRIPTION:
Rationale for treatment of uveal melanoma with sorafenib Improved understanding of the molecular pathogenesis of cancers has led to a new generation of therapeutic agents that interfere with a specific pathway critical in tumor development or progression. Although no specific genes have been linked to the pathogenesis of uveal melanoma, which significantly differs from that of cutaneous melanoma, progress has been made in identifying potential targets involved in uveal melanoma apoptosis, proliferation, invasion, metastasis, and angiogenesis. Accordingly, improvement of systemic therapy of metastatic uveal melanoma could be achieved by using molecularly targeted agents that are currently in clinical use as well as agents being tested in clinical trials. Preclinical studies suggest potential benefit of inhibitors of Bcl-2, ubiquitin-proteasome, histone deactylase, mitogen-activated protein kinase and phosphatidylinositol-3-kinase-AKT pathways, and receptor tyrosine kinases. Modifiers of adhesion molecules, matrix metalloproteinase, and angiogenic factors also have demonstrated potential benefit. (Triozzi et al, 2008).

Thus, sorafenib as oral multi-kinase inhibitor that targets the Raf/MEK/ERK signaling pathway (CRAF, BRAF, V600E BRAF) in the cell and receptor tyrosine kinases (RTKs) such as VEGFR-2, VEGFR-3, and PDGFR-ß involved in tumor cell proliferation and angiogenesis may potentially lead to a benefit for patients with metastatic uveal melanoma in terms of disease control and prolongation of survival.

In a GCP-adapted register trial approved by the ethics committee in Essen 62 patients with metastatic uveal melanoma received treatment with sorafenib on a compassionate use basis. Median overall survival was 10.8 months in patients receiving 200 mg bid sorafenib and 7.1 months in patients receiving 400 mg bid (Scheulen et al, 2011). These treatment results are encouraging for further investigation of treatment with sorafenib in patients with metastatic uveal melanoma in a randomized trial, a potential benefit of this systemic treatment is anticipated.

Rationale for selection of a randomized discontinuation trial design The randomized discontinuation trial (RDT) design , first proposed in 1975 (Amery et al, 1975) aims to assess the clinical activity of a drug while minimizing the use of placebo. All patients receive study drug for an initial run-in period, followed by random assignment of potential responders to either the study drug or the placebo (Amery et al,1975; Kopec et al,1993). RDT design provides more homogeneous study treatment groups by selecting patients with a predefined response, and allows the evaluation of a drug's clinical activity with fewer patients and increased statistical power. Thus this study design is especially useful to distinguish anticancer activity of the drug and natural history of the underlying disease (Kopec et al,1993; Jain L et al, 2006; Rosner et al, 2002). As pointed out by Rosner the RDT design is a feasible phase II study design for evaluating possible activity of cytostatic anticancer agents whereas historically anticancer drug efficacy was evaluated as being cytotoxic (Rosner et al, 2002).

As laid down in section 3.2 sorafenib is an oral multi-kinase inhibitor that targets the Raf/MEK/ERK signaling pathway in the cell and receptor tyrosine kinases (RTKs) such as VEGFR-2, VEGFR-3, and PDGFR-ß involved in tumor cell proliferation and angiogenesis. The primary clinical benefit of sorafenib is expected to be disease stabilization rather than tumor shrinkage. As disease stabilization is substantially influenced by the natural disease of a disease, the RDT design was chosen in several phase II trials evaluating possible activity of sorafenib (such as Ratain et al, 2006; Eisen et al, 2006; Pacey et al, 2009) Taking into account that uveal melanoma is a rare disease with presumably unidentified prognostic factors the RDT design seems to be useful for objective evaluation of time to progression and overall survival.

The RDT design will ensure that all patients receive treatment with sorafenib for a run-in phase of 8 weeks and will receive further treatment with sorafenib if they experience response (complete response or partial response). Patients who experience tumor progression during this run-in phase will not remain in the study but may be offered alternative treatment. Patients who experience tumor stabilization (stable disease) will be randomized double-blinded to either sorafenib or placebo. Tumor response assessments will be performed every 8 weeks, in case of progression the patient will be unblinded and offered retreatment with sorafenib if he had been randomized to placebo. Thus, if the patient experiences progression, the effective maximum duration of a possible placebo application is confined to eight weeks.

Risk-benefit assessment of the treatment of patients with metastatic uveal melanoma with sorafenib Based on the rationale for treatment of patients with metastatic uveal melanoma with sorafenib and own clinical experience in a limited number of patients with metastatic uveal melanoma treated with sorafenib on a compassionate use basis (section 3.3), a potential benefit of this systemic treatment is anticipated.

Major potential side effects of the continuous oral treatment with sorafenib are hand-foot-syndrome, diarrhoea and increase in blood pressure which can effectively be reduced either by dose reduction or cessation of treatment with sorafenib in case of hand-foot-syndrome or diarrhoea or antihypertonic agents in case of increase of blood pressure.

Further on, the administration of sorafenib (oral intake) means fewer hospitalizations and thus constitutes an improvement of quality of life.

Thus, treatment with sorafenib is a potentially effective treatment of patients with metastatic uveal melanoma without serious side effects.

In case of short-term evaluation of inappropriate antitumor efficacy patients have the option for alternative treatment strategies either by intra-arterial liver perfusion with fotemustine or melphalan in case of metastatic disease confined to the liver or salvage chemotherapy. However it should be noted that these treatments do not represent established and authorized alternative treatment options. The only randomized phase III trial comparing intra-arterial hepatic fotemustine administration with intravenous systemic fotemustine with regard to overall survival as primary endpoint is still ongoing (EORTC 18021), all other experience is based on small phase II trials or individual treatments decisions as described in section 3.1. Any locoregional treatment such as surgery or intra-arterial hepatic infusion with fotemustine or mephalan requires that the patient does not suffer from disseminated metastasis of the liver or extrahepatic localisation of metastases.

Any placement of an intra-arterial catheter and to a lower extent, intravenous catheter is associated with the risks of catheter thrombosis, dislocation, catheter stenosis/obstruction or leakage.

The main serious side effects of melphalan and fotemustine are myelotoxicity with anemia, leucopenia and thrombocytopenia and the risk of developing acute leucemia, gastrointestinal toxicity with nausea, vomiting and diarrhoea, allergic reactions, alopecia, interstitial pneumonia, liver function disorders and renal function disorders.

Considering the poor prognosis of metastatic uveal melanoma and taking into account the lack of an established treatment to treat metastatic uveal melanoma, the risk-benefit relation of the study is assessed as positive. The possible benefit of achieving disease control with sorafenib outweighs the risk of possible side effects of sorafenib. Alternative treatment options are likewise further subject to investigation, have probably more serious side effects and certainly affect the quality of life far more as result of the intraarterial/intravenous infusional application in contrast to oral intake of sorafenib.

ELIGIBILITY:
Inclusion criteria:

1. Signed and dated written informed consent before the start of specific protocol procedures
2. Metastatic uveal melanoma with histological or cytological confirmation of liver metastasis
3. By means of whole body MRI documented disease according to RECIST version 1.1 with at least one unidimensional measurable lesion ≥ 10 mm
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2
5. Male or female patients ≥ 18 years of age
6. Estimated life-expectancy more than 5 months
7. Hematologic function, as follows:

   * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
   * Platelet count ≥ 100 x 109/L
   * Hemoglobin ≥ 9 g/dL
8. Renal function, as follows

   -Creatinine ≤ 1.5 x upper limit of normal (ULN)
9. Hepatic function, as follows

   * Aspartate aminotransferase (AST) ≤ 2.5 x ULN
   * Alanine aminotransferase (ALT) ≤ 2.5 x ULN
   * Total bilirubin ≤ 3 mg/dl
   * Alkaline phosphatase ≤ 4.0 x ULN
10. PT-INR/PT < 1.5 x ULN
11. Females of childbearing potential (FCBP) must have a negative pregnancy test within 7 days of the first application of study treatment and must agree to use effective contraceptive birth control measures
12. Males must agree to use barrier birth control measures (condoms) during the course of the trial.

Exclusion criteria:

1. Previous or concurrent tumor other than uveal melanoma with the exception of cervical cancer in situ, adequately treated basal cell carcinoma, superficial bladder tumors (Ta, Tis, and T1) or any curatively treated tumors > 3 years prior to enrollment
2. History of cardiac disease: congestive heart failure ≥ NYHA class 2; active coronary artery disease ([CAD], myocardial infarction more than 6 months prior to study entry is allowed), cardiac arrhythmias requiring antiarrhythmic therapy (only beta blockers or digoxin are permitted)
3. QT/QTc-interval prolongation (QTc> 450 msec) on ECG, known Long QT syndrome or known Long QT syndrome in relatives
4. Known HIV infection
5. Known chronic infection with hepatitis B or C
6. Hypokalemia, hypocalcemia, hypomagnesemia or patients under actual treatment against hypokalemia, hypocalcemia, hypomagnesemia
7. Active infection requiring systemic antibiotic/antiviral/antifungal treatment or any uncontrolled infection > Grade 2 NCI-CTCAE
8. Symptomatic brain or meningeal tumors (unless patient is > 6 months from definitive therapy, had a negative imaging study within 4 weeks of study entry and is clinically stable with respect to the tumor at the time of study enrollment)
9. Patients with seizure disorder requiring medication (such as steroids or antiepileptics)
10. History of organ allograft
11. Patients with evidence or history of bleeding diathesis
12. Thrombotic or embolic events within the last 6 months
13. Serious non-healing wound, ulcer or fracture
14. Uncontrolled arterial hypertension with systolic blood pressure >150 mm Hg and/ or diastolic blood pressure > 90 mg Hg despite optimal treatment, determined twice within one week
15. Pregnant or breast-feeding patients
16. Marked claustrophobia
17. Cardiac pacemaker, cochlea implants or other implanted metal devices, residual metal splinters
18. Known allergy to the used study drug sorafenib or to any of its excipients
19. Known hypersensitivity to gadolinium based contrast agents
20. Subject unwilling or unable to comply with study requirements
21. Substance abuse, medical, psychological or social conditions that may interfere with the patient's participation in the study or evaluation of the study results
22. Participation in any clinical study or treatment with an experimental drug or experimental therapy within 28 days prior to study enrollment or during study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2011-06; Primary Completion 2016-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | Every 8 weeks for 1 year

SECONDARY OUTCOMES:
Number of patients with adverse events | Every 8 weeks for 1 year
Overall Survival | Every 8 weeks for 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Max E. Scheulen, Prof., Principal Investigator — Universiätsklinikum Essen
Locations (3):
- Germany (3):
  - Universitätsmedizin Berlin, Charité Campus Benjamin Franklin, Berlin
  - Universitätsklinikum Erlangen, Erlangen
  - Univesitätsklinikum Essen, Essen

REFERENCES:
- [Derived] Kalkavan H, Scheulen ME, Kampgen E, Keilholz U, Heinzerling L, Lueong SS, Hlinka A, Gromke T, Ochsenreither S, Hilger RA, Grubert M, Wetter A, Guberina N, Zeschnigk M, Ferency P, Held S, Hinke A, Schuler G, Al-Ghazzawi K, Bornfeld N, Bechrakis NE, Schuler M, Bauer S, Richly H, Siveke JT. Sorafenib as first-line therapy for metastatic uveal melanoma: A multicenter, placebo-controlled randomized discontinuation study (STREAM). iScience. 2025 Nov 14;28(12):114045. doi: 10.1016/j.isci.2025.114045. eCollection 2025 Dec 19. PMID 41362626